CLINICAL TRIAL: NCT01328301
Title: Speed-dependent Treadmill Training is Effective to Improve Gait and Balance Performance in Patients With Sub-acute Stroke
Brief Title: Effect of Speed-dependent Treadmill Training in Patients With Subacute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Tung Wah Hospital (Other)
Responsible Party: Principal Investigator, Margaret Kit Yi Mak, Dr., The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mak0001
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Stroke
Keywords: gait; hemiplegia; treadmill; physiotherapy; rehabilitation
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Speed-dependent treadmill training (SDT) (Experimental): Subjects underwent short interval of walking trials with stepwise increases in the treadmill speed
  Interventions: Other: Experimental
- speed-stable treadmill training (Active Comparator): Control subjects received gait training on the treadmill with a steady speed.
  Interventions: Other: Speed-stable treadmill training

INTERVENTIONS:
Other: Experimental — For SDT training, subjects received short intervals of locomotion training with a treadmill. After walking for 30s, the subjects were given two minutes of rest. If they completed the first walking trial safely and without stumbling, the belt speed was increased by 10% on the next trial. However, if a subject failed to complete the first trial, the belt speed was decreased by 10% on the next trial. The speed of the treadmill was adjusted in each subsequent trial according to the same principle. Subjects usually completed 7-8 walking trials in one session. The belt speed was increased by a maximum of five increments within one training session.
  Other Names: Treadmill training with increasing speed
  Arms: Speed-dependent treadmill training (SDT)
Other: Speed-stable treadmill training — Subjects in the control group walked on the treadmill with the belt speed adjusted according to their fastest over-ground gait speed. There was no adjustment of the belt speed throughout the 30-minute steady-speed treadmill training session.
  Other Names: Treadmill training with steady speed
  Arms: speed-stable treadmill training

SUMMARY:
This study aimed to explore whether speed-dependent treadmill training is more effective at improving walking and balance performance than speed-stable treadmill training in patients with subacute stroke. Twenty-six patients with stroke completed 2 weeks of treadmill training. Results showed that speed-dependent treadmill training is more effective at improving walking speed and step length than speed-stable treadmill training in patients with subacute stroke.

DETAILED DESCRIPTION:
Objectives: To compare the effects of speed-dependent treadmill training (SDT) on gait and balance performance in patients with sub-acute stroke. Design: Double-blinded randomized controlled trial. Subjects: Twenty-six patients with sub-acute stroke were randomly assigned to SDT (n=13) and control (n=13) groups. Methods: Subjects in the SDT group underwent short interval of walking trials with stepwise increases in the treadmill speed, following the principles of sprint training. Control subjects received gait training on the treadmill with a steady speed (SST). Gait speed, stride length, cadence, and Berg's balance score (BBS) were recorded and analysed before and after the 10 training sessions. Results: Results of two-way repeated measures ANOVA showed significant group x time interactions for gait speed and stride length (p < 0.05). Within each subject group, there were improvements in all gait parameters and BBS (all p < 0.001) after the training program. In addition, the SDT group showed significantly larger percentage increases in gait speed (by 72.8%) and stride length (by 29.2%) than the control subjects (p < 0.02). Conclusions: SDT in patients with sub-acute stroke resulted in larger gains in gait speed and stride length compared with SST. The positive findings provide evidence for clinical practice of SDT in enhancing gait function after stroke.

ELIGIBILITY:
Inclusion Criteria:

* first episode of stroke
* within 1 month of stroke onset
* hemiparesis resulting from unilateral ischemic stroke
* Ashworth score of 0 or 1 indicating no spasticity or slight spasticity over the affected lower limb respectively
* mini-mental status examination score of ≥ 23
* the ability to walk on level ground without physical assistance and to walk on a treadmill with a minimum speed of 22.2 cm/s for 30s

Exclusion Criteria:

* neurological diseases other than stroke,
* active cardiovascular disease (i.e. American Heart Association class C or above),
* lower limb fractures
* total hip replacement
* active rheumatoid arthritis that affected their gait performance
* Patients who required assistance to ambulate before the stroke were also excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
change in Walking speed | Change in walking speed from baseline to post-treatment, an expected average of 2 weeks
change in stride length | Change in stride length from baseline to post-treatment, an expected average of 2 weeks
change in cadence | Change in cadence from baseline to post-treatment, an expected average of 2 weeks

SECONDARY OUTCOMES:
change in Berg's balance score | Change in Berg's balance score from baseline to post-treatment, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Margaret KY Mak, PhD, Principal Investigator — Department of Rehabilitation Sciences, The Hong Kong Polytechnic University
Locations (1):
- Margaret Mak, Hong Kong, Hong Kong, China